CLINICAL TRIAL: NCT01229254
Title: A Phase II, Open-label, Dose Exposure Confirmation Study to Evaluate the Pharmacokinetics and Safety and Tolerability of Betrixaban (MK-4448) in Adult Patients With Nonvalvular Atrial Fibrillation or Atrial Flutter
Brief Title: Evaluate the Pharmacokinetics and Safety of MK-4448 in Participants With Nonvalvular Atrial Fibrillation or Atrial Flutter
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 006-00
Record Dates: First submitted 2010-09-09; First posted 2010-10-27 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Betrixaban; MK-4448; nonvalvular atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Amiodarone; betrixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amiodarone (Experimental): Participants on betrixaban 30 mg and concomitant baseline amiodarone
  Interventions: Drug: Amiodarone; Drug: Betrixaban 30 mg
- Betrixaban 60 mg (Experimental): Participants with lower weights
  Interventions: Drug: Betrixaban 60 mg
- Betrixaban 90 mg (Experimental): Participants with higher weights
  Interventions: Drug: Betrixaban 90 mg

INTERVENTIONS:
Drug: Amiodarone — Patients on Amiodarone
  Arms: Amiodarone
Drug: Betrixaban 60 mg — Betrixaban 60 mg once a day with food on Day 0 through Day 25
  Other Names: MK-4448
  Arms: Betrixaban 60 mg
Drug: Betrixaban 90 mg — Betrixaban 90 mg once a day with food on Day 0 through Day 25
  Other Names: MK-4448
  Arms: Betrixaban 90 mg
Drug: Betrixaban 30 mg — Betrixaban 30 mg once a day with food on Day 0 through Day 25 with concomitant amiodarone treatment.
  Other Names: MK-4448
  Arms: Amiodarone

SUMMARY:
The primary purpose of this study is to optimize drug exposure in the target population.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, participant requires long term anticoagulation for stroke prevention in atrial flutter (AF).
* Men and women ≥18 years of age.
* Participant has current non-valvular atrial fibrillation (NVAF) or AF or electrocardiogram (ECG) or Holter documentation within past 12 months.
* Participant has an international normalized ratio (INR) ≤ 2.2 at allocation (Visit 2).
* A participant who is of reproductive potential agrees to remain abstinent or use (or have their partner use) 2 acceptable methods of birth control for the duration of the study. Acceptable methods of birth control are: intrauterine device (IUD), diaphragm with spermicide, condom, vasectomy, and hormonal contraception.
* Participant understands the study procedures and risks involved with the study, and voluntarily agree to participate by giving written informed consent.

Exclusion Criteria:

General

* Participant is currently participating in another drug study or has received an investigational drug within 30 days prior to enrollment.
* Participant is a woman who is pregnant, lactating or of child-bearing potential who refuses to use a medically acceptable form of contraception throughout the study.
* Participant has a body weight less than 40 kg (88 lbs) or greater than 200 kg (440 lbs).
* Participant routinely consumes more than 2 alcoholic drinks per day (average >14 alcoholic drinks per week) or greater than 5 drinks within 2 hours on occasion.

Prohibited Medical Conditions

* Participant has any condition or situation which, in the opinion of the investigator, might pose a risk to the participant or interfere with participation in the study.
* Conditions associated with an increased risk of bleeding Active bleeding.
* Conditions other than AF that require chronic anticoagulation.
* Severe aortic and mitral valvular disease requiring surgical intervention.
* Previous known history of coagulopathy (e.g.: Factor V Leiden, Protein C Deficiency, Protein S Deficiency, Antiphospholipid Syndrome, etc.).
* Active infective endocarditis.
* Participant has history of familial long QT interval (the QT interval is the portion of an electrocardiogram (ECG) between the onset of the Q wave and the end of the T wave, representing the total time for ventricular depolarization and repolarization) syndrome or prolonged Bazett-corrected QT interval (QTcB) (males > 470 msec; females >480 msec) at baseline as measured on a 12-lead ECG.
* Participant has serious pulmonary, hepatic, metabolic, gastrointestinal, central nervous system (CNS) or psychiatric disease, end-stage disease states, or any other disease that could interfere with the conduct or validity of the study or compromise participant safety.
* Participant has a history of malignancy ≤ 5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer (melanoma, leukemia, lymphoma and myeloproliferative disorders of any duration are excluded).
* Participant has a history of mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy.
* Participant has reversible causes of atrial fibrillation (i.e.: cardiac surgery, pulmonary embolism, untreated hyperthyroidism).
* Participant is to undergo pulmonary vein isolation or surgery for treatment of AF.
* Participant had a severe, disabling stroke within the previous 6 months, any stroke within the previous 14 days, thromboembolism within previous 30 days or a transient ischemic attack (TIA) within 3 days prior to Visit 1.
* Participant requires renal replacement therapies (hemo- or peritoneal dialysis).
* Participant has any of a list of defined laboratory abnormalities.

Prohibited Medications

* Anti-platelet agents other than aspirin within 10 days prior to Visit 1 (excluding maintenance dose clopidogrel, prasugrel or ticlopidine) or fibrinolytic agents within 30 days prior to Visit 1.
* Aspirin greater than 162 mg/day.
* Daily non-steroidal anti-inflammatory drug (NSAID) use.
* Dronedarone, verapamil or ketoconazole.
* Vitamin K antagonists (VKA) or other anticoagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 9Sep10 & 22Apr11, 189 patients were enrolled by 68 study centers in 2 countries (USA, Canada). Patients were enrolled to 1 of 3 treatment groups (betrixaban once daily 30, 60 or 90 mg) based on weight or use of amiodarone at screening. The study had an initial pharmacokinetics (PK) phase of 4 weeks and a safety extension phase of 20 weeks.
Pre-assignment Details: Patients weighing < 80 kg received daily betrixaban 60 mg, patients weighing ≥ 80 kg received daily betrixaban 90 mg, and patients on amiodarone at screening, regardless of weight, received daily betrixaban 30 mg. 241 patients were screened for study participation. Of these patients, 189 were enrolled and received at least 1 dose of study drug.
Groups:
- Betrixaban 30 mg (+Amiodarone): Betrixaban 30 mg once daily for at least 4 weeks and up to 24 weeks for patients taking amiodarone
- Betrixaban 60 mg (<80 kg): Betrixaban 60 mg once daily for at least 4 weeks and up to 24 weeks
- Betrixaban 90 mg (≥80 kg): Betrixaban 90 mg once daily for at least 4 weeks and up to 24 weeks
Period: Overall Study
Arm/Group | Betrixaban 30 mg (+Amiodarone) | Betrixaban 60 mg (<80 kg) | Betrixaban 90 mg (≥80 kg)
Started | 42 | 74 | 73
Completed | 27 | 58 | 61
Not Completed | 15 | 16 | 12
Not completed — Not Continuing Into Safety Extension | 3 | 1 | 1
Not completed — Adverse Event | 4 | 5 | 3
Not completed — Lost to Follow-up | 3 | 0 | 1
Not completed — Physician Decision | 0 | 3 | 0
Not completed — Protocol Violation | 4 | 6 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Non-compliance with Study Drug | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients who took at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Betrixaban 30 mg (+Amiodarone) | Betrixaban 60 mg (<80 kg) | Betrixaban 90 mg (≥80 kg) | Total
Number analyzed (Participants) | 42 | 74 | 73 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (9.87) | 77.1 (7.12) | 71.2 (9.21) | 73.8 (8.98)
Age, Customized [Count of Participants; unit: Participants]
  <75 years | 23 | 24 | 46 | 93
  >=75 years | 19 | 50 | 27 | 96
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 46 | 16 | 81
  Male | 23 | 28 | 57 | 108

OUTCOME MEASURES:

1. Primary Outcome: Steady-state C12 hr on Days 14, 18, and 21 After Weight-based Dosing
Description: Betrixaban PK concentration at 12 hr on Days 14, 18, and 21 in low and high weight groups
Time Frame: Days 14, 18, and 21 of the PK period
Population: Per protocol analysis set, which includes all allocated patients who received at least one dose of study treatment and who were ≥ 90% compliant with study treatment, took study treatment within 24 hours prior to steadystate blood sampling, had at least two post steady-state blood samples collected, and not on amiodarone.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Betrixaban 30 mg (+Amiodarone) | Betrixaban 60 mg (<80 kg) | Betrixaban 90 mg (≥80 kg)
Number analyzed (Participants) | 0 | 68 | 69
ng/mL |  | 7.870 [6.654 to 9.307] | 10.517 [8.903 to 12.423]
Statistical Analysis 1: Comparison: Betrixaban 60 mg (<80 kg); Compared to Betrixaban 90 mg (≥80 kg); Test type: Equivalence — If the 90% confidence interval was within the pre-specified bounds of [0.66, 1.50], the hypothesis of similarity between lower weight and higher weight groups was supported; Ratio of geometric least-squares means = 0.748, 90% CI 2-sided [0.591 to 0.948]

2. Secondary Outcome: Steady-state C12 hr on Days 14, 18, and 21 After Weight and Amiodarone-based Dosing
Description: Betrixaban PK concentration at 12 hr on Days 14, 18, and 21 in amiodarone, low and high weight groups
Time Frame: Days 14, 18, and 21 of the PK period
Population: Full Analysis Set population, which includes all patients who received at least one dose of study treatment within 24 hours prior to steady-state (SS) blood sampling, were ≥ 90% compliant with treatment, and had at least one post SS sample. The endpoint was to summarize the SS C12 hr concentration across treatments and time points as a single arm.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Betrixaban: Betrixaban 30 mg once daily for patients taking amiodarone, plus Betrixaban 60 mg once daily, plus Betrixaban 90 mg once daily, all for at least 4 weeks and up to 24 weeks
Arm/Group | Betrixaban
Number analyzed (Participants) | 172
ng/mL | 9.498 [8.586 to 10.507]

ADVERSE EVENTS:
Time Frame: Maximum of 24 weeks
Description: Incidence of serious adverse events by system organ class
Arm/Group | Betrixaban 30 mg (+Amiodarone) | Betrixaban 60 mg (<80 kg) | Betrixaban 90 mg (≥80 kg)
Serious Adverse Events (participants affected / at risk) | 6/42 | 13/74 | 6/73
Other Adverse Events (participants affected / at risk) | 18/42 | 34/74 | 35/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Betrixaban 30 mg (+Amiodarone) (N=42) | Betrixaban 60 mg (<80 kg) (N=74) | Betrixaban 90 mg (≥80 kg) (N=73)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Betrixaban 30 mg (+Amiodarone) (N=42) | Betrixaban 60 mg (<80 kg) (N=74) | Betrixaban 90 mg (≥80 kg) (N=73)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 6
Dizziness (Nervous system disorders) | 0 | 9 | 5
Fatigue (General disorders) | 3 | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 5
Oedema peripheral (General disorders) | 3 | 3 | 5
Nausea (Gastrointestinal disorders) | 3 | 2 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4
Nasopharyngitis (Infections and infestations) | 3 | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 4 | 7 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 3 | 1
Urinary tract infection (Infections and infestations) | 2 | 9 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 4 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Due to multiple studies, centers and countries this may vary.